CLINICAL TRIAL: NCT00396591
Title: A Multicenter, Open-label, Single-arm Study of the Efficacy and Safety of Intravenous AVE0005 (VEGF Trap) Administered Every 2 Weeks in Advanced Ovarian Cancer Patients With Recurrent Symptomatic Malignant Ascites
Brief Title: AVE0005 (VEGF Trap) in Patients With Recurrent Symptomatic Malignant Ascites
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARD6772; EUDRACT: 2006-000604-16
Record Dates: First submitted 2006-11-06; First posted 2006-11-07 (Estimated); Results first posted 2013-01-10 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2011-07

CONDITIONS: Ovarian Neoplasms
Keywords: Ovarian cancer; malignant ascites; angiogenesis; angiogenesis inhibition; VEGF-Trap fusion recombinant protein
MeSH Terms: conditions — Ovarian Neoplasms | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aflibercept (Experimental): Participants with advanced ovarian epithelial cancer (including fallopian tube and primary peritoneal adenocarcinoma) treated with Aflibercept every 2 weeks until a criterion for treatment discontinuation was met
  Interventions: Drug: Aflibercept (ziv-aflibercept, AVE0005, VEGF trap, ZALTRAP®)

INTERVENTIONS:
Drug: Aflibercept (ziv-aflibercept, AVE0005, VEGF trap, ZALTRAP®) — 4.0 mg/kg administered intravenously (IV) once every 2 weeks

SUMMARY:
The primary objective of this study was to compare the time between paracenteses before and after administration of Aflibercept (ziv-aflibercept, AVE0005, VEGF trap, ZALTRAP®) in ovarian cancer participants with symptomatic malignant ascites.

The secondary objectives were to further assess efficacy and safety of Aflibercept treatment, and the exploratory objectives were to assess pharmacokinetics, immunogenicity and health-related quality of life.

DETAILED DESCRIPTION:
The study consisted of:

* A 30-day screening phase prior to Day 1
* Day 1 registration and pre-treatment paracentesis
* Aflibercept administration within 1-day of registration
* Two-week study treatment cycles (for efficacy data, the cut-off date was 6 months post-registration
* A 60-day post-treatment follow-up phase

During the study, participants were treated with Aflibercept study treatment through the duration of the study unless they met one the following criteria for discontinuation:

* Participant (or legal representative) chose to withdraw from treatment
* The investigator or sponsor thought that continuation of the study would be detrimental to the participants well-being
* Participant had intercurrent illness that prevented further administration of investigational product (IP)
* Participant had more than 2 IP dose reductions
* Participant had unacceptable adverse events (AEs)
* Participant had arterial thromboembolic events, including cerebrovascular accidents, myocardial infarctions, transient ischemic attacks, new onset angina, or worsening of preexisting angina
* Participant required surgical intervention for intestinal obstruction or gastrointestinal perforation

ELIGIBILITY:
Participants that met the following criteria were eligible.

Inclusion Criteria:

* Symptomatic malignant ascites resulting from advanced ovarian epithelial cancer (including fallopian tube and primary peritoneal adenocarcinoma) that required at least 3 previous therapeutic paracenteses at a frequency of 1 to 4 paracenteses per month for management.
* Platinum resistant disease defined by relapse or progression of disease during or after treatment, or drug intolerance.
* Topotecan- and/or liposomal doxorubicin-resistant disease defined by relapse or progression of disease during or after treatment, or drug intolerance.

Exclusion Criteria:

* Peritoneovenous or other type of shunt that was placed for the management of ascites
* Prior treatment with a VEGF or VEGF receptor inhibitor
* Uncontrolled hypertension

The above information is not intended to contain all considerations relevant to participation in a clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ICD, Study Director — Sanofi
Locations (3):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Bromma, Sweden

REFERENCES:
- [Derived] Colombo N, Mangili G, Mammoliti S, Kalling M, Tholander B, Sternas L, Buzenet G, Chamberlain D. A phase II study of aflibercept in patients with advanced epithelial ovarian cancer and symptomatic malignant ascites. Gynecol Oncol. 2012 Apr;125(1):42-7. doi: 10.1016/j.ygyno.2011.11.021. Epub 2011 Nov 21. PMID 22112608

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 17 participants were screened for this study, of which 16 participants were enrolled.
Groups:
- Aflibercept: Participants with advanced ovarian epithelial cancer treated with 4.0 mg/kg Aflibercept every 2 weeks until a criterion for treatment discontinuation was met
Period: Overall Study
Arm/Group | Aflibercept
Started | 16
Completed | 0
Not Completed | 16
Not completed — Disease Progression | 13
Not completed — Adverse Event | 2
Not completed — Participant request | 1

BASELINE CHARACTERISTICS:
Arm/Group | Aflibercept
Number analyzed (Participants) | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 59.3 (8.9)
Age, Customized [Number; unit: participants]
  <65 years | 11
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 16
Primary tumor site - Ovaries [Number; unit: Participants] | 16
Time since initial cancer diagnosis [Mean (Standard Deviation); unit: Years] | 2.8 (1.7)
Histology [Number; unit: Participants]
  Serous | 9
  Endometrioid | 3
  Clear cell (mesonephroid) | 1
  Other | 1
  Missing data | 2
Histology grade [Number; unit: Participants]
  Unknown | 5
  Moderately differentiated | 1
  Poorly differentiated | 10
Prior anticancer surgeries, [Number; unit: Participants]
  No | 1
  Yes | 15
Baseline interval of paracentesis [Mean (Standard Deviation); unit: days] — Average of the two paracentesis intervals prior to the Day 1 paracentesis before registration.
  days | 16.5 (7.8)
Eastern Cooperative Oncology Group (ECOG) performance status score [Number; unit: participants] — The ECOG score assesses how the disease affects a participant's daily living abilities. It ranges from 0-5, with 0 being the best and 5 being the worst outcome. "0" reflects a fully active participant, able to carry on all pre-disease performance without restriction. "1" reflects a participant restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. "2" reflects an ambulatory participant, who is up and about more than 50% of waking hours, and capable of all self-care but unable to carry out any work activities.
  participants
    ECOG Score = 0 | 3
    ECOG Score = 1 | 10
    ECOG Score = 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Repeat Paracentesis Response (RPR)
Description: RPR was defined as at least a two-fold increase in the time to repeat paracentesis (TRP) as compared to the average duration of the 2 intervals between the 3 most recent paracenteses prior to study registration (ie, the baseline interval of paracentesis).
  Percentage of participants with a repeat paracentesis response were the number of participants with RPR / number of total participants * 100.
Time Frame: up to 2 years post-registration
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Aflibercept
Number analyzed (Participants) | 16
percentage of participants | 62.5 [35.43 to 84.80]

2. Secondary Outcome: Time to Repeat Paracentesis (TRP)
Description: TRP is the number of days between the date of registration and the date of the first postregistration paracentesis. Median TRP was estimated from Kaplan-Meier curves. For participants who did not undergo a postregistration paracentesis while on study, TRP was censored at the end of the treatment period (last dose + 1 cycle), at the last visit known without repeat paracentesis, at 6 months postregistration, or at death, whichever was earlier.
Time Frame: up to 6 months from registration
Population: All participants were analyzed. 8 had one or more paracentesis events. Participants with no paracentesis events were censored at the end of the treatment period (last dose + 1 cycle).
Measure: Median (95% Confidence Interval); unit: days
Units Other Than Participants: Paracentesis (>/= 1 per participant)
Arm/Group | Aflibercept
Number analyzed (Participants) | 16
Number analyzed (Paracentesis (>/= 1 per participant)) | 8
days | 76.0 [64.0 to 178.0]

3. Secondary Outcome: 60-day Frequency of Paracentesis (FOP)
Description: FOP was the total number of paracenteses performed within the first 60 days postregistration. For participants who had withdrawn after registration but prior to the 60-day cutoff date, the withdrawal would have been regarded as a paracentesis event and the 60-day FOP normalized and calculated as the nearest integer of the value corresponding to 60 × number of paracenteses / x, where x represents the number of days on study.
Time Frame: up to 60 days post-registration
Measure: Mean (Standard Deviation); unit: paracenteses
Arm/Group | Aflibercept
Number analyzed (Participants) | 16
paracenteses | 1.5 (1.6)

4. Secondary Outcome: Progression-free Survival (PFS) Time
Description: According to the Response Evaluation Criteria in Solid Tumors [RECIST], progression was at least a 20% increase in the sum of the longest diameter (LD) of tumors, compared to smallest sum LD recorded since treatment started, or the appearance of one or more new tumors.
  PFS time was interval from the date of registration to the date of tumor progression or death from any cause, whichever was earlier. Median PFS time was estimated from Kaplan-Meier Plots.
  If participants were alive and progression-free at 6 months postregistration, they were censored for PFS.
Time Frame: up to 6 months post-registration
Population: Participants with a PFS event (tumor progression or death) were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Aflibercept
Number analyzed (Participants) | 12
days | 59.5 [41.0 to 83.0]

5. Secondary Outcome: Overall Survival (OS) Time
Description: OS time was the time interval between the date of registration to the date of death from any cause. Median OS was estimated from Kaplan-Meier curves. Participants who died after efficacy data cutoff date (6 months postregistration) were censored at the data cutoff date.
Time Frame: up to 6 months post-registration
Population: All participants were analyzed. 5 participants who died after efficacy data cutoff date (6 months postregistration) were censored at the data cutoff date.
Measure: Median (95% Confidence Interval); unit: days
Units Other Than Participants: Events (Death)
Arm/Group | Aflibercept
Number analyzed (Participants) | 16
Number analyzed (Events (Death)) | 11
days | 92.0 [58.0 to NA] — Not calculable as some participants were still alive at the cut-off date.

6. Secondary Outcome: Number of Participants With a Positive Anti-drug Antibody Response
Description: Anti-drug antibodies in participant's serum were measured using 2 different methods
  * an Enzyme Linked Immunosorbent Assay (ELISA) in which the lower limit of detection (LLOD) was 238.4 ng/mL; and
  * an Electrochemiluminescence-based, Bridging Assay in which the validated LLOD was about 5.4 ng/mL in the absence of aflibercept and about 25.2 ng/mL in the presence of 20 μg/mL of aflibercept.
  Participants with detectable anti-drug antibodies by either method were considered to have a positive anti-drug antibody response.
Time Frame: up to 60 days after the last dose of treatment
Population: Participants who received at least part of 1 dose of aflibercept and had evaluable blood samples
Measure: Number; unit: participants
Arm/Group | Aflibercept
Number analyzed (Participants) | 11
participants | 0

7. Secondary Outcome: Safety - Number of Participants With Adverse Events (AE)
Description: All AEs regardless of seriousness or relationship to study treatment, spanning from the first administration of study treatment until 60 days after the last administration of study treatment, were recorded, and followed until resolution or stabilization. The number of participants with all treatment emergent adverse events (TEAE), serious adverse events (SAE), TEAE leading to death, and TEAE leading to permanent treatment discontinuation are reported.
Time Frame: up to 60 days after last dose of treatment (approximately 2 years), or until TEAE was resolved or stabilized
Population: All participants who received at least part of 1 dose of the study treatment.
Measure: Number; unit: participants
Arm/Group | Aflibercept
Number analyzed (Participants) | 16
participants
  With at least one TEAE | 16
  With at least one serious TEAE | 15
  With a TEAE leading to death | 8
  With a TEAE resulting in discontinuation | 2

ADVERSE EVENTS:
Time Frame: From treatment initiation to January 30, 2009
Arm/Group | Aflibercept
Serious Adverse Events (participants affected / at risk) | 15/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aflibercept (N=16)
Anaemia (Blood and lymphatic system disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 5
Intestinal perforation (Gastrointestinal disorders) | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Disease progression (General disorders) | 4
General physical health deterioration (General disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aflibercept (N=16)
Anaemia (Blood and lymphatic system disorders) | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Conjunctivitis (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Oesophagitis (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 8
Asthenia (General disorders) | 5
Disease progression (General disorders) | 5
Early satiety (General disorders) | 2
Fatigue (General disorders) | 4
General physical health deterioration (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Oedema peripheral (General disorders) | 3
Pain (General disorders) | 2
Pyrexia (General disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Gastroenteritis (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Cardiac murmur (Investigations) | 1
Urine output decreased (Investigations) | 1
Urine output increased (Investigations) | 1
Weight decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 5
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Neuropathy peripheral (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from his site after a multicenter publication, or 12 months after the completion of the study by all sites. He must provide the sponsor a copy of any such publication derived from the study for review and comment at least 45 days (20 for abstracts) in advance of any submission for publication. The Sponsor may request for the publication to be delayed for a limited time, not to exceed 90 days to preserve its proprietary rights.